CLINICAL TRIAL: NCT06304272
Title: Comparison Between Drinking Water and Normal Saline in Irrigating Traumatic Wound: Noninferiority Trial
Brief Title: Comparison Between Drinking Water and Normal Saline in Irrigating Traumatic Wound
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Patan Academy of Health Sciences (Other)
Responsible Party: Principal Investigator, Ashis Shrestha, Assistant Professor, Patan Academy of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Irrigation
Record Dates: First submitted 2024-02-20; First posted 2024-03-12 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Trauma
Keywords: Traumatic Wound; Wound Infection
MeSH Terms: conditions — Wounds and Injuries; Wound Infection | interventions — Drinking Water; Saline Solution

STUDY DESIGN:
Intervention Model Description: Randomized, double blinded, parallel, non-inferiority trial
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Irrigating Traumatic Wound with Drinking Water (Experimental): In drinking water arm, acute traumatic wound will be cleaned with drinking water. Bacteriological safety of the drinking water will be ensured by testing water.
  Interventions: Procedure: Irrigating Traumatic Wound with Drinking Water
- Irrigating Traumatic Wound with Normal Saline (Experimental): In normal saline arm, acute traumatic wound will be cleaned with normal saline.
  Interventions: Procedure: Irrigating Traumatic Wound with Drinking Water

INTERVENTIONS:
Procedure: Irrigating Traumatic Wound with Drinking Water — Irrigating Traumatic Wound with Drinking Water and Normal Saline
  Other Names: Irrigating Traumatic Wound with Normal Saline

SUMMARY:
There is a controversy regarding the roles of the Normal saline and Tap water in irrigation of the wound. It has been suggested that antiseptic solution including normal saline has cytotoxic effect while tap water damages the fibroblast. There are no high level evidence to support one type of solution over other, systematic review have found no difference in wound infection between irrigation with normal saline vs tap water. There are ten randomized controlled trial comparing tap water with normal saline for irrigating wound published between 1992 to 2016. These RCT are analyzed in three systemic review and meta-analysis published on 2016, 2019, 2022, which showed that tap water and normal saline has no difference in terms of infection rate. The infection rate observed in various studies ranges from 0-11.5% in normal saline group and 0-12.6% in tap water group with no statistically significant difference.

DETAILED DESCRIPTION:
There is a controversy regarding the roles of the Normal saline and Tap water in irrigation of the wound. It has been suggested that antiseptic solution including normal saline has cytotoxic effect while tap water damages the fibroblast. There are no high level evidence to support one type of solution over other, systematic review have found no difference in wound infection between irrigation with normal saline vs tap water. There are ten randomized controlled trial comparing tap water with normal saline for irrigating wound published between 1992 to 2016. These RCT are analyzed in three systemic review and meta-analysis published on 2016, 2019, 2022, which showed that tap water and normal saline has no difference in terms of infection rate. The infection rate observed in various studies ranges from 0-11.5% in normal saline group and 0-12.6% in tap water group with no statistically significant difference.

The published study has looked into tap water which may not be equivalent to drinking water in our setup, therefore the investigators are looking into drinking water that is bacteriologically safe. Out of published RCTs there is only one done in acute traumatic wound with good sample size and study design. This study is purposed to look into acute traumatic wound with proper randomization, allocation and concealment. Moreover, this is a non-inferiority trial, therefore if it is proven that drinking water is non-inferior to normal saline then, it will be easily available modality of wound irrigation in Low-Middle-Income country like Nepal.

ELIGIBILITY:
Inclusion Criteria:

* Laceration wound presenting within 6 hours of duration
* Lacerations involving upper and lower limbs, scalps, head and neck

Exclusion Criteria:

* Lacerations involving, lips, ears, mucosal surface, perineal and peri anal region
* Punctured or penetrating wound
* Bite wounds by human or animals or snakes
* Dirty wound requiring surgical debridement
* Patient requiring irrigation of wound with more than 1 liter of fluid
* Wounds involving tendon, joint or bone
* Wound associated with open fracture
* Patient on corticosteroid, antibiotics or immunosuppressant
* Patient who are not able to come for follow-up
* Immunocompromised patient
* Patient with history of significant peripheral vascular disease

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 440 (Estimated)
Dates: Start 2024-03 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Comparison between drinking water and normal saline in irrigating traumatic wound: Noninferiority trial. | 3-7 Days
  Difference in wound infection rates between the two randomized groups. Wound evaluation was based on the following criteria
  No infection:
  1. No discharge or fever on day 3
  2. Dry and no fever on day 7 Infection
  1. Fever greater than 1000 F or pus discharge on any day 2. Erythema with serous discharge on any day

CONTACTS AND LOCATIONS:
Overall Officials: Ashis Shrestha, Fellow, Principal Investigator — Patan Academy of Health Sciences

REFERENCES:
- See also: The Effects of Wound Lavage Solutions on Canine Fibroblasts: An In Vitro Study — https://pubmed.ncbi.nlm.nih.gov/2344089/
- See also: Is tap water a safe alternative to normal saline for wound irrigation in the community setting? — https://pubmed.ncbi.nlm.nih.gov/12964289/
- See also: Water is a safe and effective alternative to sterile normal saline for wound irrigation prior to suturing: a prospective, double-blind, randomised, controlled clinical trial — https://pubmed.ncbi.nlm.nih.gov/23325896/
- See also: The effectiveness of cleansing solution for wound treatment A systematic review — https://www.redalyc.org/pdf/3882/388245833001.pdf
- See also: Comparison of wounds' infection rate between tap water and normal saline cleansing: A meta-analysis of randomised control trials — https://pubmed.ncbi.nlm.nih.gov/30191654/
- See also: Water for wound cleansing — https://pubmed.ncbi.nlm.nih.gov/36103365/
- See also: A Multicenter Comparison of Tap Water versus Sterile Saline for Wound Irrigation — https://pubmed.ncbi.nlm.nih.gov/17456554/
- See also: Injury, fatal and nonfatal: Sharp and cutting-edge wounds — https://asomef.org.co/wp-content/uploads/2020/04/Injury-Fatal-and-Nonfatal-Sharp-and-Cutting-Edge-Wounds.pdf
- See also: Wound classification — https://www.ncbi.nlm.nih.gov/books/NBK554456/